CLINICAL TRIAL: NCT06401447
Title: Medium Dose of Three Drugs (TPF) Concurrent Chemoradiotherapy Combined With PD-1 Checkpoint Inhibitor for Locally Advanced Esophageal Squamous Cell Carcinoma --Prospective, Single Center, Single Arm, Phase II Clinical Study (FUTURE-2)
Brief Title: TPF Concurrent Chemo-radiotherapy Plus Immunotherapy for Local Advanced Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Kailiang Wu, professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2810284-3
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): 1. Take one cycle of induction chemo-immunotherapy, two cycle of concurrent chemoradiotherapy 3 weeks later, one cycle of consolidation chemo-immunotherapy 1 month after radiotherapy, and then 1 year of immunotherapy.
  2. Radiotherapy: intensity modulated radiotherapy or volume modulated therapy. Modified involving field irradiation. PTV-C of 50.4Gy/28F, and PTV-G of 61.6Gy/28F with simultaneous integrated boost if no deep ulcers.
  3. Chemotherapy: paclitaxel 60mg/m2, ivgtt; cisplatin 30mg/m2, ivgtt; 5-FU 500mg/m2, ivgtt and 500mg/m2, civ 24h; calcium folinate 200mg; q3w.
  4. Immunotherapy: Sintilimab, 200mg, q3w.
  5. Probiotics: Clostridium Butyricum (MIYAIRI 588), 20mg, tid, for 1 year.
  6. Thymosin alpha-1: 1.6mg, qd, d1-5 during radiotherapy.
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Simultaneously optimizing the target, dosage, and synchronized drugs for radiotherapy.

SUMMARY:
The goal of this clinical trial is to learn if immune microenvironment modification could improve the effect of chemoradiotherapy for patients with local advanced esophageal squamous cell carcinoma. The main questions it aims to answer are:

1. Does immune microenvironment could be modified by medium dose of three drugs (paclitaxel, cisplatin, 5-FU), PD1 checkpoint inhibitor, probiotics, and thymosin α1？
2. Does induction and consolidation of PD1 checkpoint inhibitor improve the effect of chemoradiotherapy for patients with esophageal cancer?

This is a single arm study. Participants will:

1. Take one cycle of induction chemotherapy (paclitaxel, cisplatin, 5-FU) and immunotherapy (Sintilimab), two cycle of concurrent chemoradiotherapy, one cycle of consolidation chemo-immunotherapy, and then 1 year of immunotherapy.
2. Take probiotics (Clostridium Butyricum) for 1 year and thymosin alpha-1 daily during radiotherapy.

DETAILED DESCRIPTION:
Concurrent chemoradiotherapy is the standard treatment for patients with inoperable local advanced esophageal squamous cell carcinoma. However, over half of patients will relapse. How to improve effects? We focus on tumor microenvironment transformation by three drug chemotherapy, PD1 inhibitor, probiotics, and thymosin α1，and intent to improve radiosensitivity and reduce recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Sign written informed consent before implementing any trial related procedures;
2. Age range from 18 to 80 years old;
3. Stage II-III and stage IV esophageal squamous cell carcinoma with only extraregional lymph node metastasis determined by histopathology;
4. Inability to undergo surgical resection or patient refusal to undergo surgery;
5. ECOG PS 0-1;
6. Expected survival time>3 months;
7. Sufficient organ function is required for the subject to meet laboratory indicators

Exclusion Criteria:

1. After esophageal or tracheal stent implantation surgery;
2. Due to the obvious invasion of tumors into adjacent organs (arteries or trachea) of the esophageal lesion, there is a higher risk of Patients at risk of bleeding or perforation, or those who have formed fistulas;
3. Diagnosed as malignant diseases other than esophageal cancer within 3 years prior to initial administration (excluding those that have undergone curative treatment)
4. Currently participating in intervention clinical research treatment, or having received other treatments within 4 weeks prior to initial administration Researching drugs or using research instruments for treatment;
5. Previously received the following therapies: anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs, or targeting another stimulus or synergistic inhibition of T cell receptors (such as CTLA-4, OX-40, CD137) Medications;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 1 year
  From firt treatment to any disease progression or death

SECONDARY OUTCOMES:
clinical complete response | 1 month after radiotherapy
  disappear of tumor in CT and esophagography
Overall survival | 1 year
  From firt treatment to any death

CONTACTS AND LOCATIONS:
Overall Officials: Kailiang Wu, Doctor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No